CLINICAL TRIAL: NCT03054857
Title: The Effect of Dexmedetomidine Infusion on Post-operative Cognitive Function and Oxidative Stress in Patients Undergo Cardiopulmonary Bypass Machine Facilitated Elective Cardiac Surgery
Brief Title: The Effect of Dexmedetomidine Infusion on Post-operative Cognitive Function and Oxidative Stress in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wirinda Chiravanich, MD, Dr., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2558-102
Record Dates: First submitted 2016-06-01; First posted 2017-02-16 (Actual); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Oxidative Stress; Cognition Disorders
MeSH Terms: conditions — Cognition Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dex group (Experimental): After skin incision, the Dexmedetomidine group received a loading dose of 0.5 mcg/kg of Dexmedetomidine in 20 minutes followed by a continuous IV infusion at 0.4 mcg/kg/hr until the end of operation.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): The control group received a loading dose and continuous IV infusion of normal saline at the same rate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — After skin incision, the dexmedetomidine group received a loading dose of 0.5 mcg/kg of Dexmedetomidine in 20 minutes followed by a continuous IV infusion at 0.4 mcg/kg/hr until the end of operation.
  Other Names: Dex
  Arms: Dex group
Drug: Placebo — The control group received a loading dose and continuous IV infusion of normal saline at the same volume and rate as in the dexmedetomidine group
  Arms: Placebo group

SUMMARY:
Objective: The aim of this study was to determine the effect of dexmedetomidine in reducing postoperative cognitive dysfunction (POCD) in cardiac surgical patients which use cardiopulmonary bypass machine (CPB).

Materials and Methods: This study was double-blinded, randomized controlled trial. Patients scheduled for elective CPB facilitated cardiac surgery were randomly assigned in two groups, dexmedetomidine group (DEX) or control group. The cognitive tests (MoCA test and Short bless test) were done before the operation, 48 hours, and 7 days postoperatively. POCD was defined as a decline of 1SD of baseline score in any test. Arterial blood sample were analyzed for IL-6, IL-10, TNF-alpha and hs-CRP before induction (T0), after separation from CPB (T1), arrival at ICU (T2) and 24-hour after surgery (T3). Primary outcome was the incidence of POCD and the secondary outcomes were inflammatory response, other postoperative complications, ICU and hospital stay.

DETAILED DESCRIPTION:
After the patients were enrolled in the study, they were allocated into Dexmedetomidine group or control group by computer-based randomization. Patients, surgeons, anesthesiologists and researchers who performed the cognitive test were all blinded to the study groups.

General anesthesia was induced with intravenously midazolam 0.1-0.2 mg/kg and fentanyl 5-10 mcg/kg or Thiopental 3-5 mg/kg or Propofol 2 mg/kg. Patients were intubated with pancuronium 1 mg/kg or rocuronium 0.6-1 mg/kg. Anesthesia was maintained with nitrous oxide in oxygen, isoflurane, fentanyl, and pancuronium or rocuronium as required. Standard monitoring was provided including an indwelling radial artery catheter and central venous catheter. Bispectral index (BIS) monitoring was applied and maintained between 40-60 through the operation. Cerebral oximetry was monitored both sides of the brain by non-invasive oximeters at forehead area and the data were recorded.

After skin incision, the Dexmedetomidine group received a loading dose of 0.5 mcg/kg of Dexmedetomidine in 20 minutes followed by a continuous IV infusion at 0.4 mcg/kg/hr until the end of operation.The control group received a loading dose and continuous IV infusion of normal saline at the same rate.

During the cardiopulmonary bypass, mean arterial pressure was maintained at 60-80 mmHg or 20% from baseline. If hypertension was detected, Nicardipine 0.2 mg was given intravenously. Ephedrine 6 mg or norepinephrine 4 mcg were given within 5 minutes and repeated every 5 minutes if hypotension was presented. Atropine 0.6 mg was administered for bradycardia (heart rate less than 50 beats per minute). After the operation, patients were transferred to Cardio-thoracic intensive care unit and received standard postoperative cardiac surgery care.

2 neuropsychological tests were used to evaluate patients' cognitive function; Montreal Cognitive Assessment (MoCA) and Short blessed test (SBT). These tests were chosen by King Chulalongkorn Memorial Hospital's psychiatrist based on previous studies and the statement consensus on assessment of neurobehavioral outcomes after cardiac surgery published in 1995. All patients were evaluated their cognitive function for 3 points of time, 1st time was at preoperative period (T1), 2nd time was at 48 hours postoperatively (T2) and the last one was at 7 days postoperatively or the day at discharge from the hospital (T3). POCD was defined as a decline of 1 standard deviation (1SD) of baseline score in any test.

Blood samples were taken through the radial artery catheter, and sampling times were chosen as follows: before the induction of anaesthesia (T0); after separated from CPB (T1); arrival at intensive care unit (ICU) (T2); 24 hr after surgery (T3). Plasma Tissue Necrotic Factor-Alpha (TNF-α), Interleukin-6 (IL-6) and Interleukin-10 (IL-10) levels were measured by Magnetic Luminex Performance Assay. High sensitivity C-reactive protein (CRP) level were also measured by nephelometry.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion Criteria:

* patients who were allergy to medication in the research regimen
* preoperative left ventricular ejection fraction less than 30%
* body mass index more than 35 kg/m2
* preoperative mean arterial pressure less than 60 mmHg
* preoperative heart rate less than 45/min
* patients with impaired renal function (serum creatinine more than 1.5 mg/dl in female and 2 mg/dl in male)
* active liver disease, and who had history of symptomatic cerebrovascular disease
* psychiatric problem and other neurological diseases
* patients who cannot read

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dex Group | Placebo Group
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dex Group | Placebo Group | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.43 (13.077) | 52.72 (10.975) | 52.08 (12.017)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 26 | 32 | 58
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 49 | 50 | 99
Weight [Mean (Standard Deviation); unit: kilograms] | 60.88 (12.5) | 62.69 (11.81) | 61.794 (12.128)
BMI [Mean (Standard Deviation); unit: Kilograms per metre square] | 23.08 (3.09) | 26.19 (19.21) | 24.65 (13.8424)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage of left ventricular ejection] | 62.26 (11.53) | 63.27 (11.55) | 62.7717 (11.48959)
Serum Creatinine [Mean (Standard Deviation); unit: miligram per decilitre] | 0.94 (0.24) | 0.95 (0.27) | 0.9445 (0.25329)
Operation type [Count of Participants; unit: Participants]
  CABG | 13 | 18 | 31
  Single valve surgery | 25 | 19 | 44
  Multiple valve surgery | 6 | 12 | 18
  CABG with valve surgery | 5 | 1 | 6
Operative Time [Mean (Standard Deviation); unit: minutes] | 301.73 (87.70) | 309.28 (79.97) | 305.55 (83.541)
Cardiopulmonary Bypass Time [Mean (Standard Deviation); unit: minutes] | 120.59 (41.52) | 132.34 (46.55) | 126.53 (44.299)
Aortic Cross-clamp Time [Mean (Standard Deviation); unit: minutes] | 92.69 (34.03) | 99.88 (38.38) | 96.32 (36.287)
Diabetes Mellitus [Count of Participants; unit: Participants] | 6 | 10 | 16
Hypertension [Count of Participants; unit: Participants] | 22 | 28 | 50
Atrial fibrillation [Count of Participants; unit: Participants] | 12 | 13 | 25
Baseline Montreal Cognitive Assessment scores (0-30 points) [Mean (Standard Deviation); unit: points] — Montreal Cognitive Assessment (MoCA) is a screening test for assessment of multiple aspects of cognitive function including, attention, concentration, executive function, memory, language, calculation, visuospatial ability and orientation. MoCA score ranges from 0 to 30. Score more than 25 will be defined as normal cognitive function.
  points | 22.84 (4.464) | 22.88 (3.707) | 22.86 (4.078)
Baseline Short Blessed Test score (0-28 points) [Mean (Standard Deviation); unit: points] — Short Blessed Test (SBT) is a screening test for detecting cognitive change in the aspects of memory and concentration. SBT score ranges from 0 to 28. Score less than 4 will be defined as normal cognitive function.
  points | 4.98 (4.922) | 5.30 (5.754) | 5.14 (5.334)

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants With Postoperative Cognitive Dysfunction (POCD)
Description: POCD was defined as a decline of 1 standard-deviation (1SD) of baseline score in either MoCA test or short bless test.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dex Group | Placebo Group
Number analyzed (Participants) | 49 | 50
Participants | 12 | 8
Statistical Analysis 1: Comparison: Dex Group vs Placebo Group; Test type: Superiority; p = 0.289, Chi-squared; Risk Ratio (RR) = 1.532, 95% CI 2-sided [0.689 to 3.406]

2. Primary Outcome: Number of Participants With Postoperative Cognitive Dysfunction (POCD)
Description: POCD was defined as a decline of 1SD of baseline score in either MoCA test or short bless test.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dex Group | Placebo Group
Number analyzed (Participants) | 49 | 50
Participants | 7 | 6
Statistical Analysis 1: Comparison: Dex Group vs Placebo Group; Test type: Superiority; p = 0.636, Chi-squared; Risk Ratio (RR) = 1.329, 95% CI 2-sided [0.409 to 4.319]

3. Secondary Outcome: Number of Participants With Postoperative Complications
Description: Neurological complication, Delirium, dysrhythmia, death
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dex Group | Placebo Group
Number analyzed (Participants) | 49 | 50
Participants
  Postoperative delirium | 0 | 1
  Embolic Stroke | 0 | 1

4. Secondary Outcome: Hospital Stay in Days
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dex Group | Placebo Group
Number analyzed (Participants) | 49 | 50
days | 9.367 (3.604) | 10.42 (4.248)
Statistical Analysis 1: Comparison: Dex Group vs Placebo Group; Test type: Superiority; p = 0.187, t-test, 2 sided; Mean Difference (Final Values) = -1.053, 95% CI 2-sided [-2.626 to 0.52], Standard Deviation 0.792

5. Secondary Outcome: ICU Stay in Hours
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dex Group | Placebo Group
Number analyzed (Participants) | 49 | 50
hours | 33.79 (36.43) | 38.44 (39.17)
Statistical Analysis 1: Comparison: Dex Group vs Placebo Group; Test type: Superiority; p = 0.543, t-test, 2 sided; Mean Difference (Final Values) = -4.644, 95% CI 2-sided [-19.74 to 10.45], Standard Deviation 7.606

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Dex Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/50
Other Adverse Events (participants affected / at risk) | 13/49 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dex Group (N=49) | Placebo Group (N=50)
Cerebrovascular events (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dex Group (N=49) | Placebo Group (N=50)
dysrhythmia (Cardiac disorders) | 13 (13) | 11 (11)

LIMITATIONS AND CAVEATS:
Some missing data of postoperative neurocognitive assessment score leading to inconclusive results of some participants Low incidence of POCD in our samples leading to less reliable results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No